CLINICAL TRIAL: NCT00108017
Title: Randomized, Multicenter, Dbl-Masked, Parallel Study Evaluating the 24 Hr. Diurnal Ocular Hypotensive Effect of 2% Dorzolamide Hydrochloride/0.5% Timolol Maleate Combo. Ophthalmic Sol. in Patients w/ Open Angle Glaucoma or Ocular Hypertension
Brief Title: Comparison of the Effects of Two Glaucoma Drugs Over 24 Hours (0507A-137)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0507A-137; 2005_021
Record Dates: First submitted 2005-04-12; First posted 2005-04-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Ocular hypertension (excessive pressure in the eye)
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — dorzolamide; Timolol

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0507A, dorzolamide hydrochloride (+) timolol maleate
Drug: Comparator: timolol maleate
Drug: Duration of Treatment: Part 1) 6 wk timolol maleate run in
Drug: Part 2) 6 wk washout pd Part 3) two 8 wk active tx pds

SUMMARY:
This study is comparing 2 medications for glaucoma and how effective they are at controlling glaucoma over the course of an entire day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma or ocular hypertension

Exclusion Criteria:

* Other eye conditions
* Poor vision
* Recent eye surgery
* Use of contact lenses
* Nursing or pregnant women
* Use of some other selected medications
* Drug or alcohol abuse
* Asthma
* Slow heart beat
* Allergy or previous reaction to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2005-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
24 hour diurnal IOP reduction after 8 weeks of treatment | After 8 weeks of treatment

SECONDARY OUTCOMES:
IOP reduction a) from baseline at 6 weeks; b) comparison with timolol; c) comparison day versus night | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Feldman RM, Stewart RH, Stewart WC, Jia G, Smugar SS, Galet VA. 24-hour control of intraocular pressure with 2% dorzolamide/0.5% timolol fixed-combination ophthalmic solution in open-angle glaucoma. Curr Med Res Opin. 2008 Aug;24(8):2403-12. doi: 10.1185/03007990802243366. Epub 2008 Jul 14. PMID 18627642
- [Background] Olander KW, Galet VA, Jia G, Smugar SS, Stewart WC. Relationship between visual field severity and response to fixed combination dorzolamide/timolol or timolol alone. J Ocul Pharmacol Ther. 2009 Aug;25(4):357-64. doi: 10.1089/jop.2008.0104. PMID 19441888